CLINICAL TRIAL: NCT06913868
Title: Efficacy of a Consensus-Based Physiotherapy Approach Compared to Standardized Usual Care for the Management of Fibromyalgia: A Multicenter Randomized Controlled Trial
Brief Title: Consensus-Based vs. Standardized Physiotherapy for Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NociP-RCT-001
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Fibromyalgia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consensus-Based Physiotherapy (Experimental): Participants in this arm will receive a physiotherapy program based on the Delphi consensus recommendations of Baroni et al. (2023), tailored for individuals with fibromyalgia. This includes pain neuroscience education (approximately 20 minutes per session), tailored exercise therapy (aerobic, strengthening, and sensorimotor exercises with progressive exposure), and emphasis on self-efficacy and coping strategies. The program will be delivered by certified physical therapists trained in the consensus approach. Sessions will be 1-2 times per week for 8 weeks (60 minutes each), with a home exercise program (20 minutes, 3 times per week).
  Interventions: Behavioral: Consensus-Based Physiotherapy Program
- Usual Physiotherapy Care (Active Comparator): Participants in this arm will receive standard physiotherapy care for fibromyalgia as typically provided in outpatient settings. This may include manual therapy, home exercise prescription, and general pain education, but without the structured modules or specific emphasis on the Delphi consensus recommendations. The program will be delivered by certified physical therapists. Sessions will be 1-2 times per week for 8 weeks (60 minutes each), with a home exercise program (20 minutes, 3 times per week).
  Interventions: Behavioral: Standardized Physiotherapy Care

INTERVENTIONS:
Behavioral: Consensus-Based Physiotherapy Program — Physiotherapy for fibromyalgia (Baroni et al., 2023 Delphi consensus). Includes pain neuroscience education (PNE), tailored aerobic, strengthening, and sensorimotor exercises (graded exposure), and self-management strategies. 8-week program: 1-2 sessions/week (60 min) + home exercise (20 min, 3x/week). Therapist training and fidelity monitoring.Pain Neuroscience Education (PNE): Approximately 20 minutes per session, focusing on explaining the neurobiology of pain in fibromyalgia, emphasizing central sensitization mechanisms, and reconceptualizing pain as an output of the brain rather than solely a marker of tissue damage. PNE aims to reduce threat value associated with pain and improve understanding of pain fluctuations.
  Arms: Consensus-Based Physiotherapy
Behavioral: Standardized Physiotherapy Care — Standardized physiotherapy for fibromyalgia. Includes general exercise (aerobic, stretching), manual therapy (within guidelines), and basic pain education (excluding PNE). 8-week program: 1-2 sessions/week (60 min) + home exercise (20 min, 3x/week). Therapist training and fidelity monitoring.
  Arms: Usual Physiotherapy Care

SUMMARY:
This study compares a new, consensus-based physiotherapy program to standard physiotherapy for people with fibromyalgia. The new program uses recommendations from experts, including education about pain, personalized exercise, and strategies to improve coping skills. We will measure how much pain people have, how well they can function, and their beliefs about pain. The goal is to see if the new program is better than standard care at reducing pain and improving function in individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

Age: Adults (≥ 18 years of age).

Diagnosis: Diagnosis of fibromyalgia according to the 2016 Revisions to the 2010/2011 Fibromyalgia Diagnostic Criteria (This is the most current and recommended criteria). This requires:

Widespread Pain Index (WPI) ≥ 7 and Symptom Severity Scale (SSS) score ≥ 5 OR WPI 3-6 and SSS score ≥ 9.

Generalized pain, defined as pain in at least 4 of 5 regions (left upper, right upper, left lower, right lower, axial).

Symptoms have been present at a similar level for at least 3 months. A diagnosis of fibromyalgia is valid irrespective of other diagnoses. A diagnosis of fibromyalgia does not exclude the presence of other clinically important illnesses.

Pain Intensity: Average pain intensity of ≥ 4/10 on the Numeric Pain Rating Scale (NPRS) over the past week. (This ensures participants have clinically significant pain).

Nociplastic Pain Features:

CSI score ≥ 40. TSK score ≥ 37. Informed Consent: Willingness and ability to provide written informed consent.

Exclusion Criteria:

Red Flags: Presence of "red flags" indicating serious underlying pathology that could mimic fibromyalgia or contraindicate exercise, such as:

Unexplained weight loss. Fever or night sweats. Recent significant trauma. Neurological signs suggestive of spinal cord compression (e.g., bowel or bladder dysfunction, saddle anesthesia).

Suspected malignancy. Acute inflammatory disease. Neurological Disorders: Significant neurological deficits (e.g., multiple sclerosis, Parkinson's disease) that would interfere with participation in the study or confound outcome assessment.

Psychiatric Disorders: Uncontrolled or severe psychiatric disorders (e.g., active psychosis, severe major depression with suicidal ideation) that would preclude informed consent or adherence to the study protocol. Note: Mild to moderate, stable depression or anxiety, common in fibromyalgia, should not be an exclusion criterion.

Overlapping Pain Conditions: Presence of other significant, active pain conditions that could confound the assessment of fibromyalgia-related pain and function, such as:

Active inflammatory arthritis (e.g., rheumatoid arthritis, lupus) requiring ongoing systemic treatment.

Severe osteoarthritis requiring imminent joint replacement. Active, untreated neuropathic pain conditions (e.g., diabetic neuropathy, post-herpetic neuralgia). Note: Stable, well-managed comorbidities should not be exclusionary.

Current Pain Management: Current participation in other pain management programs or interventions that specifically overlap with the study interventions (e.g., another structured physiotherapy program, cognitive behavioral therapy specifically for pain). Note: Patients on stable doses of pain medication should not be excluded.

Exercise Contraindications: Inability to participate in exercise therapy due to medical conditions (e.g., severe cardiovascular disease, uncontrolled hypertension).

Pregnancy: Current pregnancy or planning to become pregnant during the study period. (Pregnancy can affect pain perception and exercise tolerance).

Medication Changes: Recent changes (within the past 4 weeks) in pain-related medications (e.g., opioids, antidepressants, anticonvulsants) or planned changes during the study period. Note: Stable medication regimens are acceptable.

Litigation: Current involvement in litigation related to their fibromyalgia or chronic pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2028-04-21 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Disability Index (PDI) | Baseline, 8 weeks (post-intervention)
  The PDI is a self-report questionnaire that measures the impact of pain on seven domains of daily activities: family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activities. Each domain is rated on a scale of 0-10, with higher scores indicating greater disability. The total score ranges from 0-70. The change from baseline to 8 weeks will be the primary outcome.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline, 8 weeks (post-intervention), 6-month follow-up, 12-month follow-up
  The NPRS is a single-item scale where patients rate their average pain intensity over the past week on a scale of 0-10, with 0 representing "no pain" and 10 representing "worst imaginable pain."
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 8 weeks (post-intervention), 6-month follow-up, 12-month follow-up
  The PSEQ is a 10-item questionnaire that measures a patient's confidence in their ability to perform various activities despite their pain. Each item is rated on a scale of 0-6, with higher scores indicating greater self-efficacy. The total score ranges from 0-60.
Tampa Scale of Kinesiophobia (TSK) | Baseline, 8 weeks (post-intervention), 6-month follow-up, 12-month follow-up
  The TSK is a 17-item questionnaire that measures fear of movement and (re)injury. Items are rated on a 4-point scale (strongly disagree to strongly agree), with higher scores indicating greater kinesiophobia. The total score ranges from 17-68.
Central Sensitization Inventory (CSI) | Baseline, 8 weeks (post-intervention), 6-month follow-up, 12-month follow-up
  The CSI is a 25-item questionnaire that measures the presence and severity of symptoms associated with central sensitization. Part A scores range from 0-100. Higher scores indicate a greater likelihood of central sensitization.
Patient Global Impression of Change (PGIC) | 8 weeks (post-intervention), 6-month follow-up, 12-month follow-up
  The PGIC is a single-item scale asking patients to rate their overall improvement since the start of treatment. Patients choose from a 7-point scale: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No